CLINICAL TRIAL: NCT04275674
Title: Dr. Pao-Lin Kuo (Department of Obstetrics and Gynecology
Brief Title: Inflammasome Activation and Cortisol Metabolism in Obese Women With Recurrent Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-105-481
Record Dates: First submitted 2019-10-28; First posted 2020-02-19 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood

SUMMARY:
The prevalence of obesity among women of reproductive age is increasing. Obesity represents a chronic low-grade inflammatory state and NLRP3 inflammasome plays a pivotal role in obesity-induced inflammation. Obesity is associated with an increased risk of recurrent miscarriage (RM), but the underlying mechanisms are unclear. Abnormal inflammasome activation was also identified in the endometrium of women who experienced RM. Given inflammasome activation has emerged as common pathophysiology in obesity-related disorder and RM, the investigators wonder whether inflammasome activation occurs in the uterine macrophages of obese women, and result in early reproductive failure.

DETAILED DESCRIPTION:
pending

ELIGIBILITY:
Inclusion Criteria:

All women have conceived naturally without the aid of assisted reproductive technologies

Exclusion Criteria:

N/A

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases were referred for 200 women who have experienced at least two consecutive miscarriages are recruited from outpatient clinics of our hospital, including at least 50 obese women
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Validity of inflammatory markers | 1 Day
  Use the levels of hsCRP and CA125 provides the information about inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Principal Investigator — Department of Obstetrics and Gynecology, National Cheng Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan